CLINICAL TRIAL: NCT06209229
Title: Role of Neutrophils and Electro-bioluminescence in the Therapeutic Stage of Medical Rehabilitation of Some Oncologic Diseases (Pilot Project)
Brief Title: Role of Neutrophils and Electro-bioluminescence in the Rehabilitation
Acronym: RNE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MIPO Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2
Record Dates: First submitted 2023-12-17; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Nonsmall-cell Lung Cancer
Keywords: integrative medicine; macrophages; Therapeutic Phase Of Medical Rehabilitation; Non-Small Cell Lung Cancer; sodium nucleinate; Neutrophil dysfunction test
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sodium nucleinate; Cholecalciferol; Pyridoxine; Quercetin

STUDY DESIGN:
Intervention Model Description: Simon's two-stage plan will be used (Simon R (1989). Controlled Clinical Trials 10: 1-10.). The first stage will test the Null Hypothesis that the true response rate is [p0=0.4] will be tested against the one-sided alternative hypothesis. In the first stage, [n0=16] patients will be recruited. If these [n1=34] patients have [r1=17] or fewer responses, the study will be stopped. Otherwise, [n - n1=39-34=5] additional patients will be accrued, totaling [n=39]. In the second step, the Null Hypothesis will be rejected if [r2 + 1= 20+1] or more responses are observed in [n=39] patients. This plan yields a Type I error rate [Type I error rate=0.05] and power [w=0.8] when the true response rate is [p1=0.6]. Patients will be followed up for 1 year
Masking Description: Independent sequential randomization of patients admitted over short periods of time into treatment groups will be conducted.
  Study participants will be recruited as patients present to the clinic, up to a maximum of 12 patients per week.
  Each patient included in the study will be assigned an ordinal number sequentially according to a table of a random sequence.
  For the purpose of blinding, the number will be assigned by the registrar of the admission department and will not be further involved in the study.
  The intake nurse and the researcher will not know the patient's chart except for the assigned number.
  The physician performing the examination and prescribing therapy will not know the results of the functional assessment of blood and GFR.
  The results will be entered into the subject's chart at the end of the course of treatment and supplemented by a follow-up examination after 12 months.
  Blinded follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- natirium nucleonate (Experimental): * Calcitriol- 5000 units in the morning before meals every other day 21 days and the next 3 weeks after the end of therapy.
  * Magnesium (in the form of lactate dihydrate) 470 mg + pyridoxine (in the form of hydrochloride) 5 mg - take orally 3 tablets per meter square of body surface area, in the evening 2 hours before bedtime, 21 days and the next 3 weeks after the end of therapy.
  * Quercetin from onion juice - take orally 1000 mg in the morning before meals, 21 days, as well as the next 3 weeks after the end of therapy.
  * sodium oligodinucleatide orally at the rate of 2 tablets under the tongue per meter square of body surface, in the morning 15 minutes before meals every other day, a total of 5 times (1, 3, 5, 7 , 9 day from the beginning of therapy), then after 21 days to repeat the course for 3 months.
  * Spray natirium nucleonate 4 doses in the morning on the hyoid, suck, do not swallow for 3-5 minutes, once every 4 days for 21 days.
  Interventions: Biological: sodium nucleinate

INTERVENTIONS:
Biological: sodium nucleinate — * Calcitriol- 5000 units in the morning before meals every other day 21 days and the next 3 weeks after the end of therapy.
  * Magnesium (in the form of lactate dihydrate) 470 mg + pyridoxine (in the form of hydrochloride) 5 mg - take orally 3 tablets per meter square of body surface area, in the evening 2 hours before bedtime, 21 days and the next 3 weeks after the end of therapy.
  * Quercetin from onion juice - take orally 1000 mg in the morning before meals, 21 days, as well as the next 3 weeks after the end of therapy.
  * sodium oligodinucleatide orally at the rate of 2 tablets under the tongue per meter square of body surface, in the morning 15 minutes before meals every other day, a total of 5 times (1, 3, 5, 7 , 9 day from the beginning of therapy), then after 21 days to repeat the course for 3 months.
  * Spray natirium nucleonate 4 doses in the morning on the hyoid, suck, do not swallow for 3-5 minutes, once every 4 days for 21 days.
  Other Names: cholecalciferol; pyridoxine hydrochloride; quercetin; magnesium lactate dihydrate

SUMMARY:
The clinical study is to find out the effect of a course of immunomodulatory drugs and detoxification scheme on finger bioelectroluminescence and neutrophil function and their correlation with changes in quality of life and life expectancy in patients with malignant diseases against the background of restorative treatment and rehabilitation.

Questions:

1. does the quality of life of patients with lung cancer change with the use of a course of immunomodulatory drugs and detoxification scheme?
2. does phagocytosis function, liposomal activity, mitochondrial function of neutrophils change against the background of the course?
3. does bioluminescence of fingers of hands change against the background of the course of immunotherapy? Participants will take Calcitreol capsules, Magnesium B-6 capsules, products containing quercetin flavonoids, Naderin (sodium deoxeribonucleate) daily for 21 days. before the course, after the course and after one year they will answer the QLQ-LC13, WHOQOL BREF, L.H. Garkavi adaptation self-assessment questionnaire and give blood for laboratory analysis of neutrophil function assessment.

DETAILED DESCRIPTION:
Every year, 36,000 new cases of oncology are detected in Kazakhstan, and 14,150 people (39.3%) die from oncology in Kazakhstan each year. The lowest five-year survival rate for patients with lung cancer is 12.6%. Today, an important criterion in choosing a treatment method for oncologic diseases is the level of quality of life corresponding to the treatment performed. To assess this level, special questionnaires and scales are also developed, for example, QLQ-C30 (the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 version 3.0), which appeared thanks to the separation and expansion of the GHRQL (global health-related quality of life) questionnaire. In addition to quality of life, it is very important to improve life expectancy by increasing the adaptive reserves of the organism and preventing complications. To achieve this goal it is necessary to conduct oncologic rehabilitation and course reconstructive therapy for patients with lung cancer with prevention of fiborosis development. To assess the quality of life in dynamics, it is necessary to interview patients using international questionnaires. And for objective assessment of changes in adaptation reserves it is planned to check the effectiveness of the method of functional assessment of neutrophils, bioelectroluminescence in comparison with the generally recognized neutrophil/lymphocyte index. Important in the work is the mutual control of the obtained clinical indicators with the patient's experience and his assessment of changes in the quality of life on the background of the received therapy. The expected result of the study is an increase in the average annual survival rate of patients and improved quality of life. Creation of a responsive health care system to the needs of patients.

Scientific novelty: previously such studies have not been conducted in Kazakhstan.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis Non-small cell lung cancer (histologically verified)
* Must be able to swallow tablets
* Detected for the first time
* Presence of all fingers and toes
* Patient must give their informed and signed consent
* Patient must be insured or have a health insurance plan.
* Clinically stable patients regardless of disease type.
* Absence of cognitive impairment; since the protocol provides for a clinical interview covering in particular his/her quality of life

Exclusion Criteria:

* Decompensated forms of cancer (decompensation statuses of vital organs (pulmonary, cardiac, hepatic, renal, intestinal insufficiency);
* Clinical diagnosis other types of cancer, secondary tumors and lung metastases;
* Postoperative condition for lung tumor resection;
* Patient belongs to a vulnerable group;
* Patients with severe cognitive impairment;
* Tuberculosis of any localization in the active phase and in the anamnesis;
* Severe and decompensated course of endocrine diseases, including diabetes mellitus;
* Autoimmune diseases;
* Pregnancy and lactation period;
* Prisoners;
* Active military personnel;
* People without education;
* pensioners;
* People living below the poverty line or with limited access to health services.
* Unwillingness to participate in the study.
* Patient is participating in another study
* Patient with inability to complete our protocol evaluation scales
* Patients with symptoms that compromise their level of awareness
* Insulin dependent diabetes
* Thyroid disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
scoring of completed quality-of-life tests | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Patients will be given 3 quality of life questionnaires to complete: EORTC QLQ - LC13 Lung Cancer Specific Quality of Life Questionnaire, WHOQOL Brief Quality of Life Questionnaire (WHOQOL BREF), L.H. Garkavi Adaptation Self-Efficacy Questionnaire.
survival rate | after 1 year
  Estimation of the number of patients who survived a year of rehabilitation compared to the average survival rates of public health care in the Republic of Kazakhstan
determination of stress level and adaptation reserves of the organism | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Assessment of stress level and functional adaptation reserves of the organism by bioelectrography on the GRV-camera with analysis of gas-electric photographs of the fingers of the hand in the Bio-Well program according to the following indicators: area of luminescence, normalized area, intensity of luminescence, radius of the circle inscribed in the inner oval, luminescence shape coefficient and internal noise.

SECONDARY OUTCOMES:
Total clinical morphologic blood tests | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Morphologic blood analysis with determination of the number of segmented neutrophils, basophils, monocytes and lymphocytes according to the standard of operating procedures " Total blood analysis"
A functional blood test to determine phagocytosis | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Functional blood analysis with determination of phagocytic activity of granulocytes with 1.5 μm latex and counting by a laboratory assistant of 200 cells in the ratio of stained and unstained cells in the field of lifetime light microscopy
Functional blood analysis with determination of liposomal activity of granulocytes | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Functional blood analysis with determination of liposomal activity of granulocytes by qualitative reaction to nitroblue tetrazolium and counting by a laboratory assistant of 200 cells in the ratio of stained and unstained cells in the field of lifetime light microscopy
Functional blood analysis with determination of plastic activity of granulocytes | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Functional blood analysis with determination of plastic activity of granulocytes by qualitative reaction to extra-nuclear RNA by staining with acridine orange and counting of 200 cells in the ratio of stained and unstained cells in the field of lifetime luminescent microscopy
Functional blood analysis of mitochondrial dysfunction | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Functional blood analysis with determination of mitochondrial activity of granulocytes by qualitative reaction for extra-nuclear DNA by staining with acridine orange and counting 200 cells in the ratio of stained and unstained cells in the field of lifetime luminescence microscopy by a laboratory technician
Functional blood analysis of granulocyte membrane dysfunction | Before the start of the intervention, on day 22 after the start of the intervention, and after 1 year
  Functional blood analysis of granulocyte membrane dysfunction by qualitative reaction to membrane damage by staining the cytoplasm with ethidium bromide and counting by a laboratory technician 200 cells in the ratio of stained to unstained cells in the field of lifetime luminescence microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Arai Tolemisova, PhD, Study Chair — MIPO Clinic
Locations (1):
- MIPOClinic, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No